CLINICAL TRIAL: NCT00200005
Title: Sacral Nerve Stimulation for Anal Incontinence and Bowel Control
Acronym: MDT-301
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mdt-301 November 03,1998; Mdt-301 (Nov 03, 98),; Amendment I (Dec 14, 99),; Amendment II (Jan 31, 02); Amendment III (Jul 01, 2009)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Fecal Incontinence and Constipation
Keywords: Slow transit constipation; Fecal incontinence; Constipation; Idiopathic slow transit constipation; Chronic constipation
MeSH Terms: conditions — Fecal Incontinence; Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- InterStim therapy (Experimental): Patients being treated with sacral neuromodulation with InterStim therapy.
  Interventions: Device: Type: Implantable neurostimulator; InterStim

INTERVENTIONS:
Device: Type: Implantable neurostimulator; InterStim — Treatment with InterStim Therapy: all patients meeting inclusion/exclusion criteria undergo test screening and those who have successful outcomes receive a permanent implant.
  Other Names: InterStim Model 3023; InterStim Model 3058

SUMMARY:
Multicenter European study to evaluate efficacy and safety of sacral nerve stimulation with InterStim Therapy to treat fecal incontinence or constipation

ELIGIBILITY:
140 patients (7 study groups, up to 20 implanted patients per study group)

Fecal Incontinence groups:

Main Inclusion Criteria:

* Fecal incontinence (defined as incontinence to solid or liquid stool > 1 / week);
* Failed biofeedback or medical therapy;

Groups 1 - 5 patients with:

* Group 1) Circumferentially intact external anal sphincter, no previous surgery;
* Group 2) Circumferentially intact external anal sphincter after surgical repair;
* Group 3) Rectal prolapse repaired with a rectopexy;
* Group 4) Spinal injury including disc prolapse;
* Group 5) Sigmoid or partial rectal resection with colorectal or coloanal anastomosis

Constipation groups:

Main Inclusion Criteria:

* Chronic constipation (defined as </= 2 weekly bowel movements; and/or >25% of bowel movements required straining; and/or >25% of bowel movements patient did not feel empty afterwards) with symptoms more than 1 year
* Failed biofeedback or medical therapy;

Groups 6 - 7 patients with:

* Group 6) Idiopathic slow transit constipation as proven on colonic transit studies;
* Group 7) Normal colonic transit studies but chronic constipation due to either pelvic floor dysfunction or disordered defecation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 1998-11; Primary Completion 2006-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
FI - number of FI episodes per week and/or number of days with FI per week. Constipation - number of bowel movements per week; &/or decrease defecations requiring straining; &/or decrease defecations where there was incomplete emptying | Annually

SECONDARY OUTCOMES:
FI-number of days with staining/week;urgency with continent bowel movements; Improvement in QOL;* Improvement in anal canal pressure. Constipation - Improvement in Wexner constipation score; QOL. | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Matzel, MD, Principal Investigator — University Hospital Erlangen- Erlangen, Germany; Michael A Kamm, MD, Principal Investigator — St. Vincent's Hospital- Melbourne, Australia. Former: St. Mark's Hospital, London, U.K.; Cor Baeten, MD, Principal Investigator — Maastricht University Hospital- The Netherlands; John Christiansen, MD, Principal Investigator — Herlev Hospital- Copenhagen, Denmark; Anders Mellgren, MD, Principal Investigator — Danderyd Hospital- Stockholm, Sweden; Harald Rosen, MD, Principal Investigator — Danube Hospital/SMZ-Ost- Vienna, Austria; Albert Navarro, MD, Principal Investigator — Hospital Mutua de Terrassa- Terrassa, Spain; Robert Madoff, MD, Principal Investigator — University of Minnesota- Minneapolis, USA; Carolynne Vaizey, MD, Principal Investigator — St. Mark's Hospital- London, UK; Claes Johansson, MD, Principal Investigator — Danderyd Hospital- Stockholm, Sweden; Soren Laurberg, MD, Principal Investigator — Aarhus University Hospital
Locations (9):
- University of Minnesota, Minneapolis, Minnesota, United States
- Danube Hospital/SMZ-Ost, Vienna, Austria
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Copenhagen
- University Hospital Erlangen, Erlangen, Germany
- Maastricht University Hospital, Maastricht, Netherlands
- Hospital Mutua de Terrassa, Terrassa, Spain
- Danderyd Hospital, Stockholm, Sweden
- St. Mark's Hospital, London, United Kingdom

REFERENCES:
- [Background] Matzel KE, Stadelmaier U, Hohenfellner M, Gall FP. Electrical stimulation of sacral spinal nerves for treatment of faecal incontinence. Lancet. 1995 Oct 28;346(8983):1124-7. doi: 10.1016/s0140-6736(95)91799-3. PMID 7475602
- [Result] Matzel KE, Kamm MA, Stosser M, Baeten CG, Christiansen J, Madoff R, Mellgren A, Nicholls RJ, Rius J, Rosen H. Sacral spinal nerve stimulation for faecal incontinence: multicentre study. Lancet. 2004 Apr 17;363(9417):1270-6. doi: 10.1016/S0140-6736(04)15999-0. PMID 15094271
- [Result] Jarrett ME, Matzel KE, Stosser M, Baeten CG, Kamm MA. Sacral nerve stimulation for fecal incontinence following surgery for rectal prolapse repair: a multicenter study. Dis Colon Rectum. 2005 Jun;48(6):1243-8. doi: 10.1007/s10350-004-0919-y. PMID 15793647
- [Result] Jarrett ME, Matzel KE, Christiansen J, Baeten CG, Rosen H, Bittorf B, Stosser M, Madoff R, Kamm MA. Sacral nerve stimulation for faecal incontinence in patients with previous partial spinal injury including disc prolapse. Br J Surg. 2005 Jun;92(6):734-9. doi: 10.1002/bjs.4859. PMID 15838899
- [Result] Jarrett ME, Matzel KE, Stosser M, Christiansen J, Rosen H, Kamm MA. Sacral nerve stimulation for faecal incontinence following a rectosigmoid resection for colorectal cancer. Int J Colorectal Dis. 2005 Sep;20(5):446-51. doi: 10.1007/s00384-004-0729-7. Epub 2005 Apr 21. PMID 15843939
- [Result] Kamm MA, Dudding TC, Melenhorst J, Jarrett M, Wang Z, Buntzen S, Johansson C, Laurberg S, Rosen H, Vaizey CJ, Matzel K, Baeten C. Sacral nerve stimulation for intractable constipation. Gut. 2010 Mar;59(3):333-40. doi: 10.1136/gut.2009.187989. PMID 20207638